CLINICAL TRIAL: NCT03151889
Title: Transcutaneous Electric Nerve Stimulation (TENS) Treatment for Hipossalivation Induced by Radiotherapy
Brief Title: Eletric Stimulation for Hipossalivation Induced by Radiotherapy
Acronym: TENS_HIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Fabrício Edler Macagnan, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TENS-HIR 2017
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Hyposalivation; Electric Stimulation Therapy; Head and Neck Neoplasm; Radiotherapy
MeSH Terms: conditions — Xerostomia; Head and Neck Neoplasms | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENS Group (Experimental): TENS Group: Pre-test evaluations (Clinic Conditions; Live Quality; Salivary Flux); TENS treatments (50Hz / pulse duration of 250 ms / high intensities tolerated / continuously for 20 minutes / 2 sessions a week / 4 weeks / total of the 8 TENS sessions) and Post-test evaluations.
  Interventions: Device: TENS
- Control Group (No Intervention): Control Group: Pre-test evaluations (Clinic Conditions; Live Quality; Salivary Flux) and Post-test evaluations.

INTERVENTIONS:
Device: TENS — TENS Group: Pre-test evaluations (Clinic Conditions; Live Quality; Salivary Flux); TENS treatments (50Hz / pulse duration of 250 ms / high intensities tolerated / continuously for 20 minutes / 2 sessions a week / 4 weeks / total of the 8 TENS sessions) and Post-test evaluations.
  Arms: TENS Group

SUMMARY:
Currently, cancer is a disease of high incidence, already considered a public health problem. Among the most prevalent are head and neck neoplasms, and depending on the location and extent of the lesion, the treatments are surgery, chemotherapy and / or radiotherapy that have a great impact on the quality of life. Radiation therapy is a frequently chosen treatment, and depending on the dose of radiation, causes changes such as hyposalivation. There are techniques for salivary flow stimulation, however, most of the options involve the use of medications, which limits administration to part of the patients. Transcutaneous electric nerve stimulation (TENS) is an alternative that has been used to stimulate salivary flow, however there is a limited number of studies that have tested this technique after radiotherapy. The aim of this study was to verify the effect of TENS in increasing the salivary flow of individuals receiving radiotherapy to treat tumors of the head and neck. The sample will have 80 patients randomly divided into two groups: TENS group and Control group. In both groups, a quality of life questionnaire (UW-QOL) will be applied and a speech-language assessment will be performed. The hypothesis of this research is that TENS is effective in increasing the amount of saliva. Secondary outcomes involve the evaluation of the effect of this technique on the quality of life, mainly in the questions: speech, chewing, saliva and deglutition.

DETAILED DESCRIPTION:
The sample will have 80 patients randomly divided into two groups: 1) TENS group; 2) control group. A quality of life questionnaire (UW-QOL) will be applied and a speech-language assessment will be performed. The hypothesis of this research is that TENS increasing the amount of saliva. Secondary outcomes involve the evaluation of the effect of this technique on the quality of life, mainly in the questions: speech, chewing, saliva and deglutition.

ELIGIBILITY:
Inclusion Criteria:

Starts radiotherapy treatment without previous hipossalivation

The inclusion criteria according to information contained in electronic medical records and referred by the participants are:

* Patients undergoing oncological follow-up for the treatment of head and neck cancer at Santa Rita Hospital through radiotherapy;
* Have completed radiotherapy for at least 90 days;
* Do not present a history of carcinogenic lesion in the salivary glands (sublingual, submandibular and parotid);
* Do not present oral history of oral cancer;
* Have not undergone cervical emptying level I;

Exclusion Criteria:

Intolerance to the TENS

The exclusion criteria are:

* No xerostomia;

  • Severe dysphagia;
* Stimulated salivary flow volume greater than 1.5 ml / minute;
* Use of glandular protective substances or salivary stimulants during the period of data collection;
* Use of a pacemaker or any other device that prevents electrical stimulation;
* Being pregnant;
* Unavailability of time to participate in the study (2x / week for one month);
* Excessive absences during treatment (> 30% of total sessions).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Salivary Flow | five minutes
  Salivary flow per minute (ml)

SECONDARY OUTCOMES:
Impact of the Quality of Life. | 30 days
  Questionarie University Washington

CONTACTS AND LOCATIONS:
Locations (1):
- Fabricio Edler Macagnan, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Santos FB, Vasconcelos-Raposo JJ, Figueiredo Mdo C. Correlation between symptoms and course duration of upper aerodigestive tract cancer at early and advanced stages. Braz J Otorhinolaryngol. 2013 Nov-Dec;79(6):673-80. doi: 10.5935/1808-8694.20130125. PMID 24474477
- [Result] Langendijk JA. New developments in radiotherapy of head and neck cancer: higher precision with less patient discomfort? Radiother Oncol. 2007 Oct;85(1):1-6. doi: 10.1016/j.radonc.2007.07.019. Epub 2007 Sep 12. No abstract available. PMID 17854932
- [Result] Longman LP, McCracken CF, Higham SM, Field EA. The clinical assessment of oral dryness is a significant predictor of salivary gland hypofunction. Oral Dis. 2000 Nov;6(6):366-70. doi: 10.1111/j.1601-0825.2000.tb00128.x. PMID 11355268
- [Result] Malpani BL, Jaiswar RK, Samuel AM. Noninvasive scintigraphic method to quantify unstimulated secretions from individual salivary glands. Auris Nasus Larynx. 1999 Oct;26(4):453-6. doi: 10.1016/s0385-8146(99)00026-7. PMID 10530742
- [Result] Andrews N, Griffiths C. Dental complications of head and neck radiotherapy: Part 1. Aust Dent J. 2001 Jun;46(2):88-94. doi: 10.1111/j.1834-7819.2001.tb00562.x. PMID 11491236
- [Result] Alajbeg I, Falcao DP, Tran SD, Martin-Granizo R, Lafaurie GI, Matranga D, Pejda S, Vuletic L, Mantilla R, Leal SC, Bezerra AC, Menard HA, Kimoto S, Pan S, Maniegas L, Krushinski CA, Melilli D, Campisi G, Paderni C, Mendoza GR, Yepes JF, Lindh L, Koray M, Mumcu G, Elad S, Zeevi I, Barrios BC, Lopez Sanchez RM, Lassauzay C, Fromentin O, Beiski BZ, Strietzel FP, Konttinen YT, Wolff A, Zunt SL. Intraoral electrostimulator for xerostomia relief: a long-term, multicenter, open-label, uncontrolled, clinical trial. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Jun;113(6):773-81. doi: 10.1016/j.oooo.2012.01.012. PMID 22668705
- [Result] Almeida JP, Kowalski LP. Pilocarpine used to treat xerostomia in patients submitted to radioactive iodine therapy: a pilot study. Braz J Otorhinolaryngol. 2010 Sep-Oct;76(5):659-62. doi: 10.1590/S1808-86942010000500021. PMID 20963353
- [Result] Lakshman AR, Babu GS, Rao S. Evaluation of effect of transcutaneous electrical nerve stimulation on salivary flow rate in radiation induced xerostomia patients: a pilot study. J Cancer Res Ther. 2015 Jan-Mar;11(1):229-33. doi: 10.4103/0973-1482.138008. PMID 25879367
- [Result] Strietzel FP, Lafaurie GI, Mendoza GR, Alajbeg I, Pejda S, Vuletic L, Mantilla R, Falcao DP, Leal SC, Bezerra AC, Tran SD, Menard HA, Kimoto S, Pan S, Martin-Granizo RA, Lozano ML, Zunt SL, Krushinski CA, Melilli D, Campisi G, Paderni C, Dolce S, Yepes JF, Lindh L, Koray M, Mumcu G, Elad S, Zeevi I, Barrios BC, Lopez Sanchez RM, Beiski BZ, Wolff A, Konttinen YT. Efficacy and safety of an intraoral electrostimulation device for xerostomia relief: a multicenter, randomized trial. Arthritis Rheum. 2011 Jan;63(1):180-90. doi: 10.1002/art.27766. PMID 20882668
- [Result] Dawes C, Cross HG, Baker CG, Chebib FS. The influence of gland size on the flow rate and composition of human parotid saliva. Dent J. 1978 Jan;44(1):21-5. No abstract available. PMID 272988
- [Result] Hargitai IA, Sherman RG, Strother JM. The effects of electrostimulation on parotid saliva flow: a pilot study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Mar;99(3):316-20. doi: 10.1016/j.tripleo.2004.06.080. PMID 15716838